CLINICAL TRIAL: NCT07396441
Title: Supplementary Kelulut Honey Therapy in Juvenile Open-Angle Glaucoma: Effects on IL-6, RNFL and Dry Eye.
Acronym: HONEY-JOAG
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Hospital Raja Perempuan Zainab II, Kota Bahru, Kelantan (Unknown); Hospital Sultanah Nur Zahirah, Kuala Terengganu (Other Government); Hospital Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Thamarai Munirathinam, Doctor of Medicine (MD), Medical Officer, Prinicipal Investigator, Department of Ophthalmology,, Hospital Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMRR ID-25-00996-WFT
Record Dates: First submitted 2026-01-24; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Juvenile Open Angle Glaucoma; Dry Eye Disease (DED); Interleukin 6; Retinal Nerve Fiber Layer Thickness; HbA1c Level
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Honey group (Active Comparator): Subjects will be provided stingless bee honey packeted in sachets of 30g. They are required to consume 30gram of honey per day for a total of 90 days duration.
  Interventions: Biological: Stingless bee honey (Kelulut)
- Non-honey group (No Intervention): Subjects in this group will not receive honey. Subjects will undergo comprehensive ophthalmic examination and blood taking for measurement of serum Interleukin-6 level before and after the duration of study.

INTERVENTIONS:
Biological: Stingless bee honey (Kelulut) — Kelulut is stingless bee honey, a natural biologic product produced by stinglee bee species.
  Other Names: Kelulut
  Arms: Honey group

SUMMARY:
The goal of this clinical trial is to evaluate the effects of stingless bee honey (Kelulut honey) in juvenile open-angle glaucoma patients. The study evaluates the effects on serum Interleukin 6 level(IL-6), retinal nerve fiber layer(RNFL) thickness and dry eye-related symptoms. A total of 60 participants who meet the study criteria will be randomly assigned to one of two groups. One group will consume 30 grams of Kelulut honey daily for a period of three months, while the control group will not receive honey or a placebo. Serum IL-6 level, RNFL thickness, Tear break up time (TBUT) and Schirmer Test 1 will be done before and after 90 days. Adherence to honey consumption will be monitored using a daily diary. This study aims to provide better understanding of the potential role of Kelulut honey as a supplementary therapy in patients with juvenile open-angle glaucoma.

DETAILED DESCRIPTION:
This is a randomized clinical trial conducted at four centers in Malaysia to evaluate the effects of stingless bee honey (Kelulut honey) in patients with juvenile open-angle glaucoma (JOAG). The study aims to determine whether daily consumption of Kelulut honey affects blood inflammation levels, retinal nerve fiber layer thickness, and dry eye parameters.

Two centers are assigned to the honey treatment group, and the remaining two serve as the control "no-honey" group. Participants in the honey group will consume 30 grams of Kelulut honey daily for three months, provided in sachets. The control group will continue standard glaucoma care without honey. Compliance with honey consumption will be monitored using a printed diary. Participants who experience any allergic reaction will be advised to discontinue the honey immediately and seek medical attention.

Blood samples will be collected to measure serum interleukin-6 (IL-6) levels and transported under controlled conditions to the HUSM laboratory for analysis. All participants will undergo eye examinations including retinal nerve fiber layer imaging and assessments for dry eye disease, performed using standardized procedures before and after the 3-month intervention.

ELIGIBILITY:
Inclusion Criteria:

JOAG patients age 15 years old and above until 40 years old at the time of diagnosis Compliant to conventional treatment achieved target intraocular pressure

Exclusion Criteria:

Patients with allergy to honey or honey-based products OCT signal less than 6/10 Concurrent retinal diseases and other optic neuropathies Systemic neurodegenerative disease Systemic comorbidities such as diabetes mellitus and autoimmune diseases Patients on other honey-based products for the last 3 months Patient who consumes honey-based products during the study duration of 3 months (monitoring via honey-diary, return of the used sachet during the follow up visits) Patients on anti-oxidants, traditional medications or herbal products for the last 3 months Topical usage of steroids, systemic steroids and non-steroidal anti-inflammatory drugs.

Sepsis Compliance less than 75%.

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in the level of serum Interleukin-6 level before and after consumption of stingless bee honey for 3 months among patients with juvenile open angle glaucoma | from the enrolment to the end of study at 90 days
  Blood taking will be done to evaluate any change in the level of interleukin -6
serum Interleukin 6 level | 90 days
  Measurement of serum level of Interleukin-6

SECONDARY OUTCOMES:
Change in the retinal nerve fiber layer thickness before and after consumptio of stingless bee honey in patients with juvenile open angle glaucoma | From enrollment to the end of the treatment at 90 days
  Thickness of retinal nerve fiber layer is measured using Optical Coherence Tomography

OTHER OUTCOMES:
change in the dry eye disease parameters | From enrollment until the end of study at 90 days
  Tear break-up time and Schirmer test evaluation will be done on each subjects
Change in the level of glycated hemoglobin pre and post consumption of stingless honey kelulut | From enrollment until the completion of study at 90 days
  Measurement of glycated hemoglobin will be done

CONTACTS AND LOCATIONS:
Overall Officials: Azhany Yaakub, MD, MMed, PhD, Study Director — Universiti Sains Malaysia
Locations (4):
- Malaysia (4):
  - Hospital Raja Perempuan Zainab II, Kota Bharu, Kelantan
  - Hospital Sultan Ismail Petra, Kuala Krai, Kelantan
  - Hospital Universiti Sains Malaysia, Kubang Kerian, Kelantan
  - Hospital Sultanah Nur Zahirah, Kuala Terengganu, Terengganu

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2025-06-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT07396441/Prot_ICF_000.pdf